CLINICAL TRIAL: NCT06578728
Title: Intralesional Methotrexate Injections for the Treatment of Nail Psoriasis: an Intra-subject Randomized Controlled Trial
Brief Title: Local Methotrexate Injections for the Treatment of Nail Psoriasis
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-09026516
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Nail Psoriasis
Keywords: methotrexate; triamcinolone acetonide
MeSH Terms: interventions — Methotrexate; Triamcinolone Acetonide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Intra-subject randomized controlled trial
Who Masked: Participant
Masking Description: Patient blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Intralesional Methotrexate (Experimental): Participants receive intralesional methotrexate injections into 1 nail bed/nail matrix every 6 weeks for 3 sessions.
  Interventions: Drug: Methotrexate
- Intralesional Triamcinolone Acetonide (Active Comparator): Participants receive intralesional triamcinolone acetonide injections into 1 nail bed/nail matrix every 6 weeks for 3 sessions.
  Interventions: Drug: Triamcinolone Acetonide 10mg/mL
- Intralesional Placebo (saline) (Placebo Comparator): Participants receive intralesional saline injections into 1 nail bed/nail matrix every 6 weeks for 3 sessions.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Methotrexate — 25mg/mL intralesional injection into nail bed/nail matrix
  Arms: Intralesional Methotrexate
Drug: Triamcinolone Acetonide 10mg/mL — 10mg/mL intralesional injection into nail bed/nail matrix
  Arms: Intralesional Triamcinolone Acetonide
Drug: Saline — saline intralesional injection into nail bed/nail matrix
  Arms: Intralesional Placebo (saline)

SUMMARY:
The investigators hope to learn the efficacy of methotrexate injections for treatment of nail psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age
* Subject must have nail psoriasis that is clinically diagnosed in at least 3 fingernails

Exclusion Criteria:

* Subject with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with study evaluations or optimal participation in the study. This is including, but not limited to: immunodeficiency, onychomycosis, any other nail condition other than psoriasis, allergy to methotrexate, triamcinolone acetonide, local anesthetic, normal saline, or any other material used for procedures
* Subject who has received radiation therapy, chemotherapy, and/or immunosuppressive drugs within 6 months of study, and/or oral corticosteroids or IV methotrexate for >1 month within the 6 months of study (exception inhaled steroids);
* Subjects who use substances (medications, supplements, ect) known to significantly interact with drugs used as intervention in the study
* Subject who is pregnant, breastfeeding, or planning to get pregnant
* Subject known to have received treatment with investigational drugs or devices within 30 days prior to enrollment into this study
* Subject who is on systemic treatment for psoriasis
* Subject with baseline abnormalities in liver function tests or complete blood count
* Subjects with diagnosis of renal insufficiency or impairment
* Subject who is unwilling to abstain from any cosmetic nail treatments outside those provided by the study clinic, beyond basic nail trimming (i.e. no spa nail treatments, no nail polish use, no other topical prescription nail medication)
* Subject who is unwilling to abstain from any medical nail treatments on their nails other than the study intervention (i.e. topical steroids, antifungal creams) for the duration of the study intervention and for duration of the washout period (if applicable)
* Subject who is part of the staff personnel directly involved with this study or a family member of the investigational study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of nail dystrophy as measured by the Nail Psoriasis Severity Index | Baseline (week 0), during intervention (weeks 1, 7, 13), post-intervention (weeks 17, 37)
  Mean change from baseline of the Nail Psoriasis Severity Index, which evaluates nail psoriasis symptoms with a score of 0-8 for each nail. Scores will be collected and analyzed per nail. For each nail measured by the study, patients can have a score between 0 and 8.
  A score of 0 indicates no symptoms of nail psoriasis in the nail, and a score of 8 indicates nail psoriasis features are present in four quadrants of both the nail bed and nail matrix.
Change from baseline of nail dystrophy as measured by the Physician-Assessed Global Improvement | Baseline (week 0), during intervention (weeks 1, 7, 13), post-intervention (weeks 17, 37)
  Mean change from baseline in physician-assessed global improvement severity rating which rates each nail on a 5-point scale (rating 0 - 4) based on the presence of nail plate pitting, crumbling, onycholysis, oil-drop discoloration, or nail bed hyperkeratosis.
  A score of 0 indicates none of the listed symptoms, while a score of 4 indicates severe symptoms. Scores will be collected and analyzed per nail.

SECONDARY OUTCOMES:
Treatment-Related Adverse Events | 37 weeks
  Number of participants with either treatment-related adverse events or treatment-related side effects in each treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Shari Lipner, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Israel Englander Department of Dermatology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crowley JJ, Weinberg JM, Wu JJ, Robertson AD, Van Voorhees AS; National Psoriasis Foundation. Treatment of nail psoriasis: best practice recommendations from the Medical Board of the National Psoriasis Foundation. JAMA Dermatol. 2015 Jan;151(1):87-94. doi: 10.1001/jamadermatol.2014.2983. PMID 25471223
- [Background] de Berker D. Management of nail psoriasis. Clin Exp Dermatol. 2000 Jul;25(5):357-62. doi: 10.1046/j.1365-2230.2000.00663.x. PMID 11012585
- [Background] Baran R. [How to diagnose and treat psoriasis of the nails]. Presse Med. 2014 Nov;43(11):1251-9. doi: 10.1016/j.lpm.2014.06.011. Epub 2014 Oct 16. French. PMID 25443636
- [Background] Edwards F, de Berker D. Nail psoriasis: clinical presentation and best practice recommendations. Drugs. 2009;69(17):2351-61. doi: 10.2165/11318180-000000000-00000. PMID 19911853
- [Background] de Jong EM, Seegers BA, Gulinck MK, Boezeman JB, van de Kerkhof PC. Psoriasis of the nails associated with disability in a large number of patients: results of a recent interview with 1,728 patients. Dermatology. 1996;193(4):300-3. doi: 10.1159/000246274. PMID 8993953
- [Background] Armstrong AW, Tuong W, Love TJ, Carneiro S, Grynszpan R, Lee SS, Kavanaugh A. Treatments for nail psoriasis: a systematic review by the GRAPPA Nail Psoriasis Work Group. J Rheumatol. 2014 Nov;41(11):2306-14. doi: 10.3899/jrheum.140881. PMID 25362716
- [Background] Kivelevitch D, Frieder J, Watson I, Paek SY, Menter MA. Pharmacotherapeutic approaches for treating psoriasis in difficult-to-treat areas. Expert Opin Pharmacother. 2018 Apr;19(6):561-575. doi: 10.1080/14656566.2018.1448788. Epub 2018 Mar 22. PMID 29565192
- [Background] Rigopoulos D, Baran R, Chiheb S, Daniel CR 3rd, Di Chiacchio N, Gregoriou S, Grover C, Haneke E, Iorizzo M, Pasch M, Piraccini BM, Rich P, Richert B, Rompoti N, Rubin AI, Singal A, Starace M, Tosti A, Triantafyllopoulou I, Zaiac M. Recommendations for the definition, evaluation, and treatment of nail psoriasis in adult patients with no or mild skin psoriasis: A dermatologist and nail expert group consensus. J Am Acad Dermatol. 2019 Jul;81(1):228-240. doi: 10.1016/j.jaad.2019.01.072. Epub 2019 Feb 5. PMID 30731172
- [Background] Grover C, Daulatabad D, Singal A. Role of nail bed methotrexate injections in isolated nail psoriasis: conventional drug via an unconventional route. Clin Exp Dermatol. 2017 Jun;42(4):420-423. doi: 10.1111/ced.13087. Epub 2017 Apr 10. PMID 28397295
- [Background] Jiaravuthisan MM, Sasseville D, Vender RB, Murphy F, Muhn CY. Psoriasis of the nail: anatomy, pathology, clinical presentation, and a review of the literature on therapy. J Am Acad Dermatol. 2007 Jul;57(1):1-27. doi: 10.1016/j.jaad.2005.07.073. PMID 17572277
- [Background] Wolf R, Tur E, Brenner S. Corticosteroid-induced 'disappearing digit'. J Am Acad Dermatol. 1990 Oct;23(4 Pt 1):755-6. doi: 10.1016/s0190-9622(08)81079-1. No abstract available. PMID 2229508
- [Background] Requena L, Zamora E, Martin L. Acroatrophy secondary to long-standing applications of topical steroids. Arch Dermatol. 1990 Aug;126(8):1013-4. No abstract available. PMID 2383026
- [Background] Deffer TA, Goette DK. Distal phalangeal atrophy secondary to topical steroid therapy. Arch Dermatol. 1987 May;123(5):571-2. No abstract available. PMID 3579338
- [Background] Tosti A, Piraccini BM, Cameli N, Kokely F, Plozzer C, Cannata GE, Benelli C. Calcipotriol ointment in nail psoriasis: a controlled double-blind comparison with betamethasone dipropionate and salicylic acid. Br J Dermatol. 1998 Oct;139(4):655-9. doi: 10.1046/j.1365-2133.1998.02462.x. PMID 9892909